CLINICAL TRIAL: NCT06402591
Title: Multiple Doses Versus Single Dose of Cefazolin to Prevent Periprosthetic Joint Infection After Revision Arthroplasty: a Multicenter Open-label, Randomized Clinical Trial.
Brief Title: Results of Extended Versus Single Dose Antibiotic Prophylaxis In Orthopedic Revision Arthroplasty in Nijmegen.
Acronym: REViSION
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Sint Maartenskliniek (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NL70114.091.19
Record Dates: First submitted 2023-04-07; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Infection Prosthesis Hip and Knee; Infection, Prosthesis Related; Joint Infection; Infection, Surgical Site; Surgical Site Infection; Infection Pro
MeSH Terms: conditions — Prosthesis-Related Infections; Surgical Wound Infection | interventions — Cefazolin

STUDY DESIGN:
Intervention Model Description: randomized controled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- single dose cefazolin prophylaxis (No Intervention): prophylaxis according current guidelines single dose 2000mg cefazolin 15-30 minutes before incision
- extended cefazolin prophylaxis (Experimental): 5 days of cefazolin prophylaxis start dose 2000mg followed by 14 doses of 1000mg
  Interventions: Drug: Cefazolin

INTERVENTIONS:
Drug: Cefazolin — cefazolin extended prophylaxis 5 days (15 doses)
  Arms: extended cefazolin prophylaxis

SUMMARY:
The goal of this randomized control trial is to investigate the superiority of 5 days (extended) versus a single dose of cefazolin prophylaxis in revision arthroplasty of the hip and knee. The main question[s] it aims to answer are:

* Is an extended regimen compared to a single dose of cefazolin associated with an increased infection-free implant survival within one year after index revision arthroplasty of the hip or knee?
* What are the incidence, risk factors, treatment outcome and prognosis of surgical site infections and periprosthetic joint infection during follow-up?
* What is the safety and tolerance of the antimicrobial prophylaxis regimens used?
* What are the antimicrobial susceptibility patterns of micro-organisms causing PJI during follow-up?
* What is the patient' physical performance and satisfaction of subjects within 1 year after the index revision arthroplasty, using patient related outcome measurements (PROMS)?

[question 2] Participants will [describe the main tasks participants will be asked to do, treatments they'll be given and use bullets if it is more than 2 items]. If there is a comparison group: Researchers will compare [insert groups] to see if [insert effects].

DETAILED DESCRIPTION:
Periprosthetic joint infection (PJI) is an important complication of total joint arthroplasty of the hip and knee and occurs in 1-2% after primary arthroplasty and in 10-15% after revision arthroplasty. To prevent a PJI, peri-operative antibiotic prophylaxis is given. There's inadequate evidence for a recommendation about the optimal duration of prophylaxis, especially in revision arthroplasty. The aim of this multicenter open-label, randomized controlled trial is to investigate the superiority of 5 days (extended) versus a single dose of cefazolin prophylaxis in revision arthroplasty of the hip and knee. Patients will be recruited at the orthopedic departments of two Dutch hospitals, University Medical Center Radboudumc Nijmegen (Radboudumc) and Sint Maartenskliniek in Nijmegen (SMK). Patients will be included if they will undergo revision arthroplasty of the hip or knee, with exclusion of patients with a proven PJI at baseline. A total of 780 subjects will be randomized between 2 prophylactic strategies: A) Cefazolin at a single dose of 2 grams intravenously 15-60 minutes before incision; B) Cefazolin at a dose of 2 grams intravenously 15-60 minutes before incision, followed by cefazolin 1 gram intravenously t.i.d. until five days post-surgery. The primary endpoint is the difference in proportion of infectious-free implant survival between both groups within 1 year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older.
2. Planned revision arthroplasty of the hip or knee prosthesis (index revision arthroplasty), with revision of one or more fixed components.

Exclusion Criteria:

1. If the index revision arthroplasty has been cancelled.
2. Revision of single mobile parts only.
3. PJI on baseline, based on 'definite infection' score according to the Philadelphia consensus definition 2018
4. PJI on baseline, based on a positive culture of a single synovial fluid or tissue sample yielding a high virulence micro-organism (S. aureus, Enterobacterales, Pseudomonas spp, Acinetobacter spp, Candida spp).
5. Contraindication to cefazolin:

a. Previous allergic reaction according to the criteria in Appendix A. b. Severe kidney disease defined as eGFR <10 ml/min. f. Antimicrobial treatment within 3 days prior to index revision arthroplasty. g. Subjects who are currently enrolled in investigational immunosuppressive drug trials.

h. Subjects who are unable to provide informed consent.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 751 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Success rate of revision arthroplasty | 1 year after revision arthroplasty
  1. Implant retention during follow-up,
  2. No 'definite infection' score for PJI according to the Philadelphia consensus definition 2018 during follow-up
  3. No PJI based on positive culture of a single synovial fluid or tissue sample yielding a high virulence micro-organism (S. aureus, Enterobacteriaceae, Pseudomonas spp, Acinetobacter spp, Candida spp) during follow-up.
  4. No more than 4 consecutive weeks of systemic antimicrobial therapy for any reason during follow-up.

SECONDARY OUTCOMES:
incidence surgical site infections | 1 year after revision arthroplasty
  a. The proportion of SSI according to PREZIES (PREventie van ZIEkenhuisinfecties door Surveillance) criteria in both study groups during follow-up.
incidence periprosthetic joint infection | 1 year after revision arthroplasty
  The proportion of PJI according to Philadelphia consensus definition 2018 in both study groups during follow-up.
resistance rate of causative of SSI/PJI to cefazolin | 1 year after revision arthroplasty
  The cefazolin susceptibility of the micro-organisms causing SSI and PJI in the study groups.
The number of repeated surgeries. | 1 year after revision arthroplasty
  The number of repeated surgeries.
Reason repeated surgery | 1 year after revision arthroplasty
  The reason for repeated surgery on the affected prosthetic joint during follow-up.
adverse drug events | 1 year after revision arthroplasty
  Adverse drug events and serious adverse events.
Risk factors associated with SSI and PJI: BMI, age, age of implant before revision, | 1 year after revision arthroplasty
  Risk factors associated with SSI and PJI: BMI, age, age of implant before revision, number of previous revisions before index
Implant survival at the end of the study. | during inclusion of the study
  Implant survival at the end of the study.
Patient related outcome measurements | 1 year after revision arthroplasty
  PROMs at weeks 12 and 52

CONTACTS AND LOCATIONS:
Overall Officials: Bart-Jan Kullberg, prof. Dr, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No